CLINICAL TRIAL: NCT01993524
Title: Efficacy and Safety Assessment of prOVag Dietary Supplement in Recurrent Bacterial Vaginitis. Multi-centre, Randomized, Double-blind, Placebo-controlled Clinical Study.
Brief Title: Supplementation of Standard Antibiotic Therapy With Oral Probiotics for Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSS Biomed S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PB-DM/SBK-prOVag2-01/08
Record Dates: First submitted 2013-10-29; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Bacterial Vaginosis; Bacterial Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Experimental): At I visit standard treatment(500mg oral metronidazole twice daily for 7 days) and probiotic twice daily for 10 days. At II visit, participants were checked for signs of vaginal infection; if they were still present they were given a targeted antibiotic according to the microbiological analysis. Antibiotic was taken together with probiotic twice daily for 10 days. Participants showing positive response to metronidazole treatment on the II visit were given only the probiotic once daily for 10 days in the peri-menstrual period for the next 3 months. Participants with targeted antibiotic were to come to the visit IIbis, and if treatment was successful they were to proceed for the next 3 months in the same manner as those successfully treated with metronidazole, as described above.
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): At I visit standard treatment (500mg oral metronidazole twice daily for 7 days) and placebo twice daily for 10 days. At the II visit, participants were checked for signs of vaginal infection; if they were present they were given a targeted antibiotic according to the microbiological analysis. Antibiotic was taken together with placebo twice daily for 10 days. Participants showing positive responses to metronidazole on the II visit were given only placebo once daily for 10 days in the peri-menstrual period for the next 3 months. Participants with targeted antibiotic were to come to the visit IIbis, and if treatment was successful they were to proceed for the next 3 months in the same manner as those successfully treated with metronidazole, as described above.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: probiotic — antibiotic plus probiotic
  Arms: probiotic
Other: placebo — antibiotic plus placebo
  Arms: placebo

SUMMARY:
The purpose of this study was to determine whether supplementation of standard antibiotic therapy with oral probiotic preparation prOVag containing lactic acid bacteria influences recurrence of bacterial vaginosis/vaginitis.

DETAILED DESCRIPTION:
Bacterial vaginosis is the most common vaginal infection in women of reproductive age. This condition is caused by an overgrowth of anaerobic bacteria with concomitant reductions in Lactobacillus populations in the vagina, i.e. disruption of the vaginal microbiota. Aerobic vaginitis is related to the suppression of lactobacilli by various aerobic bacteria, mostly originating from the anal microbiota.

Previous open-label study confirmed that probiotic strains - Lactobacillus fermentum 57A, Lactobacillus plantarum 57B, and Lactobacillus gasseri 57C given orally to women with intermediate/abnormal vaginal flora and no clinical symptoms had the ability to colonize rectum and vagina and contributed to the maintenance of pH level and Nugent score. The colonisation of women with tested strains had been confirmed by microbiological and molecular methods.

The purpose of this multicentre, randomized study was to investigate whether the use of a probiotic preparation containing Lactobacillus fermentum 57A, Lactobacillus plantarum 57B, and Lactobacillus gasseri 57C together with standard treatment for bacterial vaginosis/vaginitis could reduce the recurrence rates of these conditions, as assessed using clinical and microbiological criteria, in comparison with standard treatment alone. The study took place between March 2009 and February 2012 in nine private out-patient gynaecological clinics in the Krakow area and Katowice (Silesia) in Poland. It was conducted in accordance with the original protocol and according to ICH-GCP requirements. The duration of subject's participation in the trial was approximately 5-6 months (follow-up visit included). As the trial did not concern medicinal product but the foodstuff (dietary supplement) it did not require Authority approval but was only subject to relevant Ethics Committee approval.

Women with history of recurrent bacterial vaginosis/vaginitis, aged 18 - 50 years, who complied with inclusion and exclusion criteria and who signed informed consent form were enrolled and randomized into one of the study groups.

Efficacy parameters were based on the evaluation of clinical symptoms during gynaecological examinations, as well as the determination of vaginal pH, Nugent score, total Lactobacillus counts and presence/numbers of vaginal pathogens in cultures from vaginal swabs collected at each visit. Data obtained at the third-fifth visits were compared with those obtained at the first visit. Clinical samples were transported to central laboratory for further analysis.

Safety parameters were analysed using information recorded in 'patient's diaries' throughout the study period, as well as the investigator's assessments at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form
2. Subjects aged more than or equal 18 and less than or equal 50 years
3. Women of the Caucasian race
4. Regularly menstruating premenopausal women (normal menstrual function (Eumenorrhoea) shall mean regular menstrual bleeding pattern every 28 plus/minus 10 days)
5. No irregularities identified in gynaecological examination (no pathology of reproductive organs, such as myomas, ovarian cysts)
6. Susceptibility to recurrent vaginitis and/or urinary tract infections, as well as bacterial vaginitis confirmed at visit I

Exclusion Criteria:

1. Subjects aged less than 18 and more than 50 years
2. Hypersensitivity to any ingredient of the investigational product, metronidazole or antibiotic(s).
3. Bleeding from genital tract of unknown aetiology
4. Pregnancy
5. Breastfeeding
6. Congenital and acquired immunodeficiencies
7. Diabetes
8. Mental illness
9. Neoplastic disease
10. Application of mechanical contraceptives, such as: diaphragms, intrauterine contraceptive insert (except for Mirena intrauterine device)
11. Application of NuvaRing hormonal contraceptive vaginal ring
12. Application of hormonal preparations, such as: Vagifem, Ovestin and vaginal estrogens in reproductive period
13. Application of another oral and/or vaginal probiotic at Subject qualification to the Study
14. Participation in another clinical study / less than thirty-day interval from the last clinical study
15. Mycotic vaginitis
16. Antibiotic therapy for other reasons
17. Pathology of reproductive organs (myomas, ovarian cysts, etc.)
18. Scheduled surgery or hospitalization

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 594 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduced probability of recurrent bacterial vaginosis/vaginitis. | assesed on visits III-V (assesed monthly within three months)
  Recurrence of bacterial vaginosis/vaginitis at the third-fifth visits was considered to be the study endpoint (participant's withdrawal). The reduced probability of recurrent bacterial vaginal infection, confirmed by clinical and/or microbiological symptoms, was the parameter used to assess primary efficacy.

SECONDARY OUTCOMES:
Change in vaginal pH level. | assesed monthly within five-six months
  Determination of pH level of vaginal discharge using indicator paper at each visit, comparison of the test outcome with the test result at Visit I.
Change in Nugent score level. | assesed monthly within five-six months
  Assessment according to the Nugent score at each visit; comparison of the outcomes with the assessment at Visit I.
Change in total Lactobacillus counts a in cultures from vaginal swabs. | assesed monthly within five-six months
  Total count of Lactobacillus bacteria in vaginal flora in material collected at each visit.Data obtained at the third-fifth visits were compared with those obtained at the first visit.
The time to bacterial vaginosis/vaginitis recurrence | assesed on visits III-V (assesed monthly within three months)
  The time to bacterial vaginosis/vaginitis recurrence was measured from the visit on which a participant showed no symptoms: the second visit for participants on standard metronidazole treatment and the second visit bis for participants treated with metronidazole and targeted antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Chelmicki, MD, PhD, Principal Investigator — "Polis CLINIC" Prywatna Opieka Lekarska Specjalistyczna Sp. z o.o, ul. 1-go Maja 88, 40-240 Katowice, Poland; Aleksandra M Cichonska, PhD, Study Director — IBSS Biomed S.A.

REFERENCES:
- [Derived] Heczko PB, Tomusiak A, Adamski P, Jakimiuk AJ, Stefanski G, Mikolajczyk-Cichonska A, Suda-Szczurek M, Strus M. Supplementation of standard antibiotic therapy with oral probiotics for bacterial vaginosis and aerobic vaginitis: a randomised, double-blind, placebo-controlled trial. BMC Womens Health. 2015 Dec 3;15:115. doi: 10.1186/s12905-015-0246-6. PMID 26635090